CLINICAL TRIAL: NCT05201352
Title: Multicentric Randomized Phase I/II Study to Evaluate Efficacy of Trifluridine/Tipiracil Plus XB2001 (Anti-IL-1α True Human Antibody) Versus Trifluridine/Tipiracil Plus Placebo in Metastatic Colorectal Cancer Patients After Failure of Oxaliplatin, Irinotecan, Fluoropyrimidine
Brief Title: Evaluation of Efficacy of Trifluridine/Tipiracil Plus an Anti-IL-1α True Human Antibody Versus Trifluridine/Tipiracil Plus Placebo in Metastatic Colorectal Cancer Patients After Failure of Oxaliplatin, Irinotecan, Fluoropyrimidine
Acronym: TASKIN
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004601-31
Record Dates: First submitted 2021-12-28; First posted 2022-01-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: trifluridine/tipiracil; anti-IL-1α True Human antibody; phase I/II
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; tipiracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental arm (Experimental): trifluridine/tipiracil + XB2001
  Interventions: Drug: trifluridine/tipiracil + XB2001
- Control arm (Placebo Comparator): trifluridine/tipiracil + placebo
  Interventions: Drug: trifluridine/tipiracil + placebo

INTERVENTIONS:
Drug: trifluridine/tipiracil + XB2001 — trifluridine/tipiracil every 28 days + XB2001 1000mg intravenous infusion every 2 weeks
  Arms: Experimental arm
Drug: trifluridine/tipiracil + placebo — trifluridine/tipiracil every 28 days + Placebo intravenous infusion every 2 weeks
  Arms: Control arm

SUMMARY:
Unresectable metastatic colorectal cancer (mCRC) remains an incurable disease. After failure of conventional treatments involving fluoropyrimidines, oxaliplatin and irinotecan in combination or not with biotherapies targeting EGFR and VEGF; regorafenib shows a modest improvement in overall survival. Recently, trifluridine/tipiracil has also shown efficacy in phase 3 with an overall survival of around 7 months. Trifluridine/tipiracil has become the standard of care for advanced mCRC in most western countries. However, the objective response rate remains very low and the survival gain remains moderate (+2 months). Therefore, new strategies are needed to ensure that mCRC patients who have received multiple lines of therapy can receive more effective treatments.

Based on previous clinical trials on IL-1 inhibition and our preclinical data, IL-1 inhibition may increase the efficacy of trifluridine/tipiracil. The goal is to test whether the addition of XB2001 to trifluridine/tipiracil could be synergistic.

DETAILED DESCRIPTION:
This project proposes to evaluate trifluridine/tipiracil plus XB2001 in patients with metastatic colorectal cancer previously treated with oxaliplatin, fluoropyrimidine and irinotecan in combination or not with an anti-angiogenic and an anti-EGFR for RAS Wild type tumor.

The project will consist of a randomized (1:1 ratio), double-blind, non-comparative, multi-center Phase II study with two treatment arms:

* Experimental arm: trifluridine/tipiracil + XB2001
* Control arm: trifluridine/tipiracil + placebo

ELIGIBILITY:
Inclusion Criteria:

* Male or female that must have signed a written informed consent prior to any study specific procedures
* Aged ≥ 18 years at randomization
* Patient with histologically proven metastatic colorectal cancer previously treated for metastatic disease by chemotherapy treatment including oxaliplatin, irinotecan, fluoropyrimidine, antiangiogenic (anti-VEGF: bevacizumab or aflibercept) and anti-EGFR (cetuximab or panitumumab) if indicated (MSI tumor could be included if previously pretreated with anti PD1/PDL1 therapy) n.b:
* a patient treated with oxaliplatin in a neoadjuvant/adjuvant situation with a recurrence of the disease within 6 months following the last administration is considered resistant to oxaliplatin and validates the criterion if no administration of oxaliplatin has been carried out in a metastatic disease situation.
* exception for VEGF if medically contraindicated during previous metastatic disease treatment (should be clearly documented in the disease history of the patient) it is allowed to included the patient with or without Bevacizumab.
* Have a performance status of 0 or 1 according to the WHO Easter Cooperative Oncology Group (ECOG)
* Knowledge of RAS, BRAF, Microsatellite status
* Baseline tumoral evaluation (thoraco-abdomino-pelvic computed tomography) perfromed within 21 days before randomization with at least one measurable lesion according to RECIST 1.1 criteria.
* Patient willing and able to comply with protocol for the duration of the study including: scheduled visits and exams, visits during the follow-up and treatment compliance.
* Adequat hepatic, renal and bone marrow function within the following limits:
* Total bilirubin ≤ 1,5 times the upper limit of normal (ULN) (unless documented Gilbert's syndrome);
* ASAT et ALAT ≤ 5 times ULN;
* Measured Creatinine clearance (Cockcroft and Gault) > 30 ml / min
* Absolute Neutrophil Count (ANC) > 1,5. 109 / L;
* Platelet count ≥ 150. 109 / L;
* Haemoglobin ≥ 9 g / dL (patients can be included even if they have been transfused)
* Albuminemia ≥ 30 g / L;
* Negative Hepatitis B, C and HIV serologies, or absence of active B or C hepatitis
* Urea protein, urine dipstick should be less than 2 crossese and/or 24 hour proteinuria ≤ 1g/24h
* Availability of tumor material dated less than 5 years with sufficient quantity (15 to 20 whithe slides) and quality (Good morphological conservation / Presence of tumor tissue / Histopathology consistent with the indication / More than 100 tumor cells)
* Patient must be affiliated to a social health insurance
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients (urine within 72h or serum pregnancy within 14 days prior to inclusion).
* Women of childbearing potential willing to use adequate contraception method (including the use of a mechanical method of contraception in the event of hormonal contraceptive treatment) during the treatment period and 6 months following the end of treatment.
* Male patients with a partner of childbearing potential should use effective contraception during treatment and for up to 6 months after stopping treatment.
* Normal ECG or ECG without clinically significant findings with QTcF < 470 ms.

Exclusion Criteria:

* Other concurrent malignancies the last 3 years, except adequately treated cone-biopsied in situ carcinoma (as per exemple of the cervix, basal cell, squamous cell carcinoma of the skin, low risk prostate cancer or other insitu carcinoma juged eligible according the coordinator). Patient who have had potentially curative therapy for a prior malignancy are eligible provided there has been no evidence of disease for ≥ 3 years and the risk of recurrence is considered low.
* Symptomatic brain metastases
* Estimated prognosis <3 months.
* Mutational status BRAF mutant (V600E only)
* Participation in progress, or in the 30 days preceding the first scheduled day of dosing in this study, in another therapeutic trial with an experimental molecule or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer.
* Severe unbalanced illness, underlying infection that may prevent the patient from receiving treatment. Patients with a clinically important and unresolved Grade 3 or 4 non-haematologic adverse reaction related to previous therapies. Also participant with any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Bowel obstruction or sub-obstruction or a history of inflammatory bowel disease or significant gasto intestinal disorder
* History of autoimmune or inflammatory disease or interstitial lung disease.
* Patient with congenital galactosemia, total lactase deficiency (lactose intolerance) or glucose-galactose malabsorption syndrome
* Severe arterial thromboembolic events less than 6 months before randomization
* New York Heart Association (NYHA) Class III or IV congestive heart failure, ventricular arrhythmias or uncontrolled blood pressure (defined as ≥ 160/100 mm Hg)
* Clinically significant decrease in performance status (medical records) within 2 weeks of intended first dose administration.
* -Contraindication to receive a treatment with trifluridine/tipiracil or an anti-IL-1α (XB2001 True Human antibody) and/or patient already treated by trifluridine/tipiracil, or an anti-IL-1α.
* Concomitant systemic treatment with immunotherapy, immunosuppressants, corticosteroid therapy ≥ 10 mg equivalent prednisone/prednisolone or hormone therapy: corticosteroid therapy administered chronically, immunosuppressive treatment, biotherapy administered as part of the management of an inflammatory disease (anti-TNF, anti-IL6, anti-IL1, anti PD-1, anti EGFR etc.) and live virus vaccines administered up to 14 days prior the first scheduled dose of treatement administration.
* Current pregnancy (mandatory pregnancy test at baseline for female of childbearing potential) or breastfeeding.
* Patient with any psychiatric, psychological, sociological, geographical problem or other severe concomitant disease, disorder or condition that potentially compromising the understanding of the information, the safety of the patient, the interpretation of study results or the conduct of the study compliance with the study protocol and follow-up schedule.
* Patient deprived of their liberty or under guardianship, curatorship or safeguard of justice.
* Known or suspected history of immunosuppression, including history of invasive opportunistic infections (e.g tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution. Presence or suspicion of active bacterial, fungal or viral infections, or uncontrolled fever.
* Major surgery within 2 weeks prior to randomization or have an unhealed operation wounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-10-13 (Actual); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-10-13 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of XB2001 | At the end of Cycle 1 (each cycle is 28 days)
Overall survival | 6-month

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - Centre Georges-François Leclerc, Dijon, Bourgogne-Franche-Comté
  - CHU Dijon, Dijon, Bourgogne-Franche-Comté
  - ICO Angers, Angers
  - Institut Sainte Catherine, Avignon
  - CHU Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Hospitalier Carcassonne, Carcassonne
  - CHU Estaing, Clermont-Ferrand
  - Hopital Franco-Britannique, Levallois-Perret
  - CHU Dupuytren, Limoges
  - CHU Nantes, Nantes
  - Cario-Hpca, Plérin
  - Institut Jean Godinot, Reims
  - Institut de Cancérologie de l'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fumet JD, Roussot N, Bertaut A, Limagne E, Thibaudin M, Hervieu A, Zanetta S, Borg C, Senellart H, Pernot S, Thuillier F, Carnot A, Mineur L, Chibaudel B, Touchefeu Y, Martin-Babau J, Jary M, Labourey JL, Rederstorff E, Lepage C, Ghiringhelli F. Phase I/II study of trifluridine/tipiracil plus XB2001 versus trifluridine/tipiracil in metastatic colorectal cancer. Future Oncol. 2024;20(38):3077-3085. doi: 10.1080/14796694.2024.2415280. Epub 2024 Nov 12. PMID 39530624